CLINICAL TRIAL: NCT00625599
Title: Fractures in the Elderly Population of El Salvador at Hospital Zacamil: Exploring Knowledge, Causes, Risk Factors, and Outcomes
Status: Completed | Type: Observational
Sponsor: Edward Via Virginia College of Osteopathic Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: Evcom-13
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2008-01

CONDITIONS: Osteoporosis; Fractures in the Elderly
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Salvadorian students at the Evangelical University in non-health track studies over the age of 18. The students must accept the invitation to participate along with signing the informed consent to be eligible.
  Interventions: Other: Osteoporosis Prevention Information
- 2: Patients over the age of 45 presenting to Hospital Zacamil with an acute fracture. Patients must accept the invitation to the study and sign the informed consent to be eligible.
  Interventions: Other: Osteoporosis Prevention Information

INTERVENTIONS:
Other: Osteoporosis Prevention Information — Primary investigator designed osteoporosis prevention information.

SUMMARY:
As the population's life expectancy increases, fractures among the elderly in El Salvador are also increasing. There is currently limited data specific to the incidence and cause of fractures in the elderly within developing countries, such as El Salvador. The problem of inadequate knowledge pertaining to bone health and osteoporosis among the elderly is contributing to this aging population's health issues. The purpose of this study is to investigate the incidence, prevalence, and risk factors effecting elderly patients admitted for fractures at the Hospital Zacamil in San Salvador, El Salvador. The study will also assess the current knowledge in two distinct populations on bone health and osteoporosis. The first population will be the patients over the age of 45 that present to Hospital Zacamil with acute fractures and are consulted by the department of orthopedics. The second population will consist of students at the Evangelical University over the age of 18 in non-medial track studies. All individuals will have to accept the invitation to participate in the study. In addition, educational materials will be developed on the prevention of fractures for medical professionals and for the elderly in El Salvador. The study objectives will determine incidence and prevalence of elderly fractures of patients over the age of 45 at Hospital Zacamil. Secondly, the study will look at demographic information, prevalent causes of fractures, treatment of the fractures, morbidity and mortality, and any complications that may arise in the fracture patients prior to their discharge from the hospital. Thirdly, the study will seek out the current level of knowledge on bone health, osteoporosis, and fracture prevention in the young, educated Salvadorians and patients over the age of 45 at Hospital Zacamil. Fourthly, the study will address the benefits of the information gained by use of educational materials with the patients and doctors of El Salvador.

Hypothesis One:

Fractures of the elderly at Hospital Zacamil are significantly associated with occurring at the hip, wrist, and vertebra in comparison to other fracture locations.

ELIGIBILITY:
Inclusion Criteria:

* For the student population they must be over the age of 18 and a student in non-medical track studies.
* For the patient population they must be over the age of 45 and present to Hospital Zacamil with an acute fracture.

Exclusion Criteria:

* Not accepting the invitation to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There will be two populations for this study. Hospital patients, females and males, over the age of 45 that are admitted to the department of orthopedics at the Hospital Zacamil in San Salvador, El Salvador from January 2008 to April 2008 will represent one of the populations. All patients over the age of 45 presenting to the hospital due to an acute fracture will be invited to join the study. The individual's care will not be changed negatively or positively based on whether or not the individual decides to participate in this study.
  The second population group will be the university students, females and males, over the age of 18 participating in non-medical studies at the Evangelical University in February 2009. No student will be negatively affected by not participating in this study. There will be no positive or negative influence on the student's grade or course assessment from participating or choosing not to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- El Salvador (2):
  - Evangelical University, San Salvador
  - Hospital Zacamil, San Salvador